CLINICAL TRIAL: NCT01978431
Title: Impulsivity and Stimulant Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Gustavo Angarita, Assistant Professor of Clinical Psychiatry, Yale University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1001006250; R25MH071584 (NIH)
Record Dates: First submitted 2013-10-17; First posted 2013-11-07 (Estimated); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Cocaine Dependence; Impulsivity
MeSH Terms: conditions — Cocaine-Related Disorders; Impulsive Behavior | interventions — Cocaine; Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Stimulant (Experimental): Cocaine and Methylphenidate
  Interventions: Drug: cocaine hydrochloride; Drug: methylphenidate
- Placebo (Placebo Comparator): methylphenidate
  Interventions: Drug: methylphenidate

INTERVENTIONS:
Drug: cocaine hydrochloride
  Arms: Stimulant
Drug: methylphenidate

SUMMARY:
Examine the interaction between stimulants, such as cocaine and methylphenidate, and impulsivity.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 - 50 years,
2. voluntary, written, informed consent,
3. physically healthy by medical history, physical, neurological, ECG, and laboratory examinations,
4. DSM-IV criteria for Cocaine Abuse (305.60) or Cocaine Dependence (304.20)
5. recent street cocaine use in excess of amounts to be administered in the current study,
6. intravenous and/or smoked (crack/ freebase) use,
7. positive urine toxicology screen for cocaine,
8. for females, non-lactating, no longer of child-bearing potential (or agree to practice effective contraception during the study), and a negative serum pregnancy (β-HCG) test.

Exclusion Criteria:

1. Other drug dependence (except nicotine) as determined by urine toxicology or interview
2. < 1 year of cocaine dependence,
3. a primary major DSM-IV psychiatric diagnosis (schizophrenia, bipolar disorder, etc.), unrelated to cocaine,
4. a history of significant medical (cardiovascular) or neurological illness, ie prior myocardial infarction, current active symptoms of cardiovascular disease / angina, evidence of cocaine-related cardiovascular symptoms, prior arrhythmias or need for cardiovascular resuscitation, neurovascular events such as transient ischemic attacks, stroke, and/or seizures Parameters re: elevations in vital signs are now explicitly specified under "Safety features built into our one-day self-administration paradigm).
5. current use of psychotropic and/or potentially psychoactive prescription medication,
6. seeking treatment for drug abuse/dependence (for experimental cocaine component),
7. physical or laboratory (β-HCG) evidence of pregnancy.
8. current use of any medication (prescription or over-the-counter) determined to cause potential drug interactions by the study physicians.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Mean cocaine inter-infusion interval | 3 hours
  Subjects complete three separate 60 minute long "binge" cocaine self administration sessions (low dose 8mg/70kg, medium dose 16mg/70kg, and large dose 32mg/70kg). Mean inter-infusion intervals (time between cocaine boluses) are then averaged by adding all intervals within each session and dividing by 60. Intervals during which pump access is withheld (due to increase in vital signs) will be excluded. Data on cocaine self-administration (total number of responses, infusions, and III), subjective effects, and vital signs will be checked for normality prior to analysis using Kolmogorov-Smirnov statistics and normal probability plots. The significance level for all statistical tests will be set at p<.05.

SECONDARY OUTCOMES:
Stop Signal Reaction Time (Impulsivity) | 5 years
  The Dependent measures pertinent to the effects of an acute/chronic exposure to stimulants (methylphenidate/cocaine) on measures of impulsivity will be analyzed using a mixed design ANOVA. This design will have a within subjects variable to study the effects of an acute exposure to stimulants (methylphenidate vs. placebo) and a between subjects variable to study the effects of a chronic exposure to stimulants (cocaine dependent subjects vs. healthy controls).
Inter-Temporal Choice (Impulsivity) | 5 years
  The Dependent measures pertinent to the effects of an acute/chronic exposure to stimulants (methylphenidate/cocaine) on measures of impulsivity will be analyzed using a mixed design ANOVA. This design will have a within subjects variable to study the effects of an acute exposure to stimulants (methylphenidate vs. placebo) and a between subjects variable to study the effects of a chronic exposure to stimulants (cocaine dependent subjects vs. healthy controls).

CONTACTS AND LOCATIONS:
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Kohler RJ, Zhornitsky S, Potenza MN, Yip SW, Worhunsky P, Angarita GA. Cocaine self-administration behavior is associated with subcortical and cortical morphometry measures in individuals with cocaine use disorder. Am J Drug Alcohol Abuse. 2024 May 3;50(3):345-356. doi: 10.1080/00952990.2024.2318585. Epub 2024 Mar 29. PMID 38551365